CLINICAL TRIAL: NCT03463057
Title: A Phase II Study Evaluating the Feasibility and Clinical Efficacy of Atezolizumab Consolidation Treatment in High Risk Diffuse Large B-cell Lymphoma
Brief Title: The Feasibility and Clinical Efficacy of Atezolizumab Consolidation Treatment in High Risk (IPI > 2) DLBCL
Acronym: HO151DLBCL
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stichting Hemato-Oncologie voor Volwassenen Nederland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HO151; 2017-002605-35 (EudraCT Number)
Record Dates: First submitted 2018-02-23; First posted 2018-03-13 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-10

CONDITIONS: NHL; DLBCL
MeSH Terms: interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Atezolizumab (Other): 18 cycles atezolizumab followed by 12 months of observation
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Intervention Atezolizumab starts after 6 - 8 R-CHOP induction cycles (Rituximab, Cyclophosphamide, Hydroxo-doxorubicin, Vincristine and Prednisone (R-CHOP)); 18 cycles Atezolizumab followed by 12 months of observation
  Other Names: Tecentriq; L01XC

SUMMARY:
The prognosis of Diffuse Large B cell Lymphoma (DLBCL) patients with an early relapse is dismal. Atezolizumab has shown promising activity in relapsed DLBCL patients. Toxicity data on atezolizumab are available for > 6000 patients and is manageable. The assumption of this study is that atezolizumab consolidation will result in higher disease free survival by eradicating minimal residual disease In melanoma and lung cancer consolidation immunotherapy after chemoradiotherapy has shown an increase in survival.

DETAILED DESCRIPTION:
In high risk diffuse large B-cell lymphoma (DLBCL), International Prognostic Index (IPI)-score ≥ 3 21% of patients will relapse within 2-years after completion of R-CHOP induction treatment despite achieving a complete remission. Patient relapsing within a year after R-CHOP treatment have a very poor prognosis, even after second line chemotherapy, with only 15% of patients achieving a long remission. Therefore, additional therapy in first line treatment is required for these patients. The immune checkpoint inhibitor atezolizumab is a monoclonal antibody directed against the program death ligand 1 (PDL1). The PD1 and PDL1 inhibitors have shown excellent results in relapsed Hodgkin lymphoma and promising results in relapsed B-cell non Hodgkin lymphoma. Given the acceptable toxicity profile of atezolizumab, this study examines the efficacy and toxicity of atezolizumab as consolidation treatment after R-CHOP induction in DLBCL patients at high risk of relapse.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 (inclusive) years
* Patients with a confirmed histologic diagnosis of diffuse large B-cell lymphoma (DLBCL-NOS) based upon a representative histology specimen according to the World Health Association (WHO) classification, revision 2016
* Ann Arbor stages II-IV
* WHO performance status 0 - 1
* International Prognostic Index (IPI) ≥ 3 at diagnosis
* Complete metabolic remission (Deauville 1-3) after 6-8 cycles of R-CHOP according to the Lugano criteria

Of note:

1. Rituximab may have been administered either intravenously or subcutaneously. A rituximab biosimilar may have been used when it is approved for the indication of DLBCL.
2. Patients should have received at least 6 cycles R-CHOP. Dose reductions for vincristine are allowed during R-CHOP. Dose reductions because of bone marrow toxicity are allowed but cannot exceed >15% of cumulative dose of doxorubicin and cyclophosphamide.
3. Central nervous system prophylaxis (MTX) by intrathecal therapy or IV is allowed.
4. Fludeoxyglucose Positron Emission Tomography (18F-FDG-PET) scan should have been made 4-8 weeks after last induction cycle
5. Histologically confirmed false positive EoT PET-scans are eligible.

   * Negative pregnancy test at study entry
   * Patient is willing and able use adequate contraception during and until 5 months after the last protocol treatment.
   * Patient is capable of giving a written informed consent

   Exclusion Criteria:

   Diagnosis

   • All histopathological diagnoses other than DLBCL-NOS according to the WHO classification, revision 2016, including:

   - High-grade B-cell lymphoma with a double/triple translocation with MYC, BCL2 and/or BCL6. Please note that patients with an isolated MYC translocation or an isolated BCL2 translocation or an isolated BCL-6 translocation are eligible (single hit translocation).
   * Testicular large B-cell lymphoma
   * Primary mediastinal B cell lymphoma
   * Transformed indolent lymphoma
   * Post-transplant lymphoproliferative disorder

   Organ dysfunction
   * Clinical signs of severe pulmonary dysfunction
   * Clinical signs of heart failure (New York Heart Association (NYHA) classification II-IV)
   * Symptomatic coronary artery disease or cardiac arrhythmias not well controlled with medication.
   * Myocardial infarction during the last 6 months
   * Significant renal dysfunction (serum creatinine ≥ 150 umol/l or clearance ≤ 30ml/min

   Creatinine clearance (CrCl) may be calculated by Cockcroft -Gault formula:

   CrCl = (140 - age [in years]) x weight [kg] (x 0.85 for females)/(0.815 x serum creatinine [μmol/L])

   • Inadequate hematological function: hemoglobin < 5.5 mmol/L Absolute Neutrophil Count (ANC) < 1.0x10↑9/L or platelets < 75x10↑9 /L
   * Signs or known history of bleeding disorder.
   * Significant hepatic dysfunction (total bilirubin ≥ 1.5x upper limit of normal (ULN) or transaminases ≥ 2.5 x ULN), unless related to Gilberts syndrome.
   * Clinical signs of severe cerebral dysfunction
   * Patients with a history of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant and adversely affecting compliance to study drugs
   * Major surgery within the last 4 weeks

   Known or suspected infection • Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection or any major episode of infection requiring treatment with IV antibiotics or hospitalization within 4 weeks of the start of Cycle 1. Suspected active or latent tuberculosis needs to be confirmed by positive interferon gamma (IFN-γ) release assay

   • Patients known to be Human Immuno-deficiency Virus (HIV)-positive
   * Active chronic hepatitis B or C infection
   * Administration of a live, attenuated vaccine within 4 weeks before date of registration or anticipation that such a live attenuated vaccine will be required during the study and for a period of 5 months after discontinuation of atezolizumab

   Auto-immune • Any active or history of documented autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.

   The following exceptions are allowed: Patients with autoimmune-related hypothyroidism or type 1 diabetes mellitus who are on stable treatment.
   * History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis per chest computer tomography (CT) scan at screening.
   * Patients with uncontrolled asthma or allergy, requiring systemic steroid treatment
   * Regular treatment with corticosteroids within the 4 weeks prior to date of registration, unless administered for indications other than NHL at a dose equivalent to < 30 mg/day prednisone/prednisolone

   General

   • Serious underlying medical conditions, which could impair the ability of the patient to participate in the trial (e.g. ongoing infection, uncontrolled diabetes mellitus, gastric ulcers, active autoimmune disease)

   • Current participation in another clinical trial interfering with this trial

   • History of active cancer during the past 5 years, except basal cell carcinoma of the skin, stage 0 cervical carcinoma or carcinoma in situ (for which no systemic treatment was indicated)

   • Life expectancy < 6 months

   • Any psychological, familial, sociological and geographical condition potentially hampering compliance with the study protocol and follow-up schedule

   Prior treatment
   * Prior treatment with Atezolizumab, or anti-programmed cell death protein-1 (anti PD-1) or PDL-1 antibodies.
   * Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA4 therapeutic antibodies.
   * Treatment with systemic immunostimulatory agents (including but not limited to IFN, interleukin [IL]-2) within 6 weeks or 5 half-lives of the drug, whichever is shorter, prior to Cycle 1, Day 1.
   * Treatment with systemic immunosuppressive medications, including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor (anti-TNF) agents within 2 weeks prior to date of registration; inhaled corticosteroids and mineralocorticoids are allowed.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) measured from the date of registration to relapse or death from any cause whichever comes first. | 2 year after inclusion last patient
  To evaluate the 2-year DFS for patients in complete metabolic remission after R-CHOP induction

SECONDARY OUTCOMES:
(Severe) Adverse Events and the relation of adverse events in time to the recovery of the T-cell repertoire. | 2 years after inclusion last patient
  To evaluate toxicity and assess the relation of adverse events in time to recovery of the T-cell repertoire.
Overall survival (OS), calculated from registration until death from any cause. Patients still alive or lost to follow up are censored at the last date known to be alive. | 2 years after inclusion last patient
  To evaluate the 2-year OS.
The relationship between MRD status at the end-of-induction and end-of-consolidation therapy. | 2 years after inclusion last patient
  To evaluate MRD status at the end of induction therapy, at various time points during consolidation treatment and at the end of consolidation.
The relation between MRD conversion and 2-years DFS and OS. | 2 years after inclusion last patient
  To evaluate if there is a relation between MRD conversion and 2-years DFS and OS.
The relation between the T-cell and NK cell repertoire and adverse events. | 2 years after inclusion last patient
  To evaluate the recovery of the T-cell and NK cell repertoire after induction therapy and at various time points during consolidation treatment in relation to toxicity and efficacy.

OTHER OUTCOMES:
Atezolizumab spinal fluid concentration as assessed by spinal fluid measurements will be performed in patients receiving atezolizumab. | 2 years after inclusion last patient
  To assess the crossing of the blood-brain barrier of atezolizumab by measuring atezolizumab concentrations in het cerebrospinal fluid.

CONTACTS AND LOCATIONS:
Overall Officials: M. Nijland, PhD/MD, Principal Investigator — NL-Groningen-UMCG
Locations (32):
- Belgium (5):
  - BE-Antwerpen Edegem-UZA, Antwerp
  - BE-Antwerpen-ZNASTUIVENBERG, Antwerp
  - BE-Brugge-AZBRUGGE, Bruges
  - BE-Leuven-UZLEUVEN, Leuven
  - BE-Roeselare-AZDELTA, Roeselare
- Netherlands (27):
  - NL-Den Bosch-JBZ, 's-Hertogenbosch
  - NL-Amersfoort-MEANDERMC, Amersfoort
  - NL-Amsterdam-OLVG, Amsterdam
  - NL-Amsterdam-VUMC, Amsterdam
  - NL-Apeldoorn-GELREAPELDOORN, Apeldoorn
  - NL-Breda-AMPHIA, Breda
  - NL-Delft-RDGG, Delft
  - NL-Dordrecht-ASZ, Dordrecht
  - NL-Ede-ZGV, Ede
  - NL-Eindhoven-CATHARINA, Eindhoven
  - NL-Eindhoven-MAXIMAMC, Eindhoven
  - NL-Enschede-MST, Enschede
  - NL-Groningen-UMCG, Groningen
  - NL-Hilversum-TERGOOI, Hilversum
  - NL-Hoofddorp-SPAARNEGASTHUIS, Hoofddorp
  - NL-Leeuwarden-MCL, Leeuwarden
  - NL-Leiden-LUMC, Leiden
  - NL-Maastricht-MUMC, Maastricht
  - NL-Nieuwegein-ANTONIUS, Nieuwegein
  - NL-Nijmegen-CWZ, Nijmegen
  - NL-Rotterdam-ERASMUSMC, Rotterdam
  - NL-Rotterdam-MAASSTADZIEKENHUIS, Rotterdam
  - NL-Sittard-Geleen-ZUYDERLAND, Sittard
  - NL-Den Haag-HAGA, The Hague
  - NL-Tilburg-ETZ, Tilburg
  - NL-Utrecht-UMCUTRECHT, Utrecht
  - NL-Zwolle-ISALA, Zwolle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nijland M, Issa DE, Bult JAA, Deeren D, Velders GA, Nijziel MR, Sandberg Y, Vergote V, Oosterveld M, Fijnheer R, Brouwer RE, Boersma RS, Wu K, Nieuwenhuizen L, Vermaat JSP, van Kampen RJW, Terpstra WE, Snauwaert S, van der Poel MW, de Jongh E, Durian MF, Strobbe L, Beeker A, Gadisseur A, van Rijn RS, Visser O, Doorduijn JK, Snijders TJF, Silbermann MH, de Jong D, Chamuleau M, Mous R, Jalving H, Visser-Wisselaar H, Jansen van de Bergh S, Zwezerijnen GJC, Bremer E, Brink M, Diepstra A, Chitu DA, Koene HR, Zijlstra JM. Atezolizumab consolidation in patients with high-risk diffuse large B-cell lymphoma in complete remission after R-CHOP. Blood Adv. 2025 Jul 22;9(14):3530-3539. doi: 10.1182/bloodadvances.2024015226. PMID 40249860
- See also: HOVON website — http://www.hovon.nl